CLINICAL TRIAL: NCT00905021
Title: EXTENT: Exemestane (AROMASIN®) in Combination With Sunitinib (SUTENT®) in Hormone Receptor Positive Metastatic Breast Cancer
Brief Title: Exemestane With Sunitinib (SUTENT®) in Metastatic Breast Cancer
Acronym: EXTENT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew support
Sponsor: Baylor Breast Care Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Mothaffar Rimawi, Medical Director, Baylor Breast Care Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H 24786 / EXTENT
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer; Metastatic; Hormone Receptor Positive
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — exemestane; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exemestane plus Sutent (Experimental): All patients enrolled on the study will receive treatment as follows:
  1. Exemestane 25 mg by mouth every day.
  2. Sunitinib 37.5 mg by mouth every day.
  Interventions: Drug: Exemestane; Drug: Sutent

INTERVENTIONS:
Drug: Exemestane — Exemestane 25 mg by mouth every day.
  Other Names: Aromasin
Drug: Sutent — Sunitinib 37.5 mg by mouth every day.
  Other Names: (Sunitinib)

SUMMARY:
The investigators want to find out if the treatments used in this study are helpful to patients that are diagnosed with hormone receptor positive metastatic breast cancer. The investigators want to also look at any side effects that could happen while patients are on the study treatments. The investigators want to see if there are any changes that could show us if your cancer is responding to the study treatments.

DETAILED DESCRIPTION:
The study design is a phase II design. Eligible patients will undergo staging work up and start treatment. Every 28-day period (4 weeks) will count as a cycle. Medical evaluations will be performed every 4 weeks and staging work up will be repeated every 12 weeks.

The primary objective of the study is to assess progression free survival (PFS) of treatment with exemestane and sunitinib in post¬menopausal subjects with hormone receptor positive (ER-positive and/or PR-positive) unresectable locally advanced or metastatic breast cancer subjects who have progressed on prior hormonal treatment.

In addition we want to:

1. Obtain assessments of overall response rate (ORR), clinical benefit rate (CBR), and overall survival (OS).
2. Determine the safety and tolerability of the combination regimen.
3. Study molecular changes in tissue biopsies, circulating tumor cells (CTCs), and circulating endothelial cells (CECs), and explore associations with treatment response and resistance.

1. Blood samples will be drawn for enumeration and profiling of circulating tumor cells and circulating endothelial cells at study entry (prior to starting study medications), four weeks after starting study medications, twelve weeks after starting study medications and at disease progression. These samples will be strongly encouraged but the patients may decline any or all of them without impacting their eligibility or continuation on the study.

2. If the patient participating on the study has an easily accessible breast mass or metastatic lesion (e.g. lymphadenopathy, skin metastasis, chest wall metastasis), a core needle or punch biopsy will be obtained at study entry (prior to starting study medications), four weeks after starting study medications, and at disease progression. These biopsies will be strongly encouraged but the patients may decline any or all of them without impacting their eligibility or continuation on the study.

ELIGIBILITY:
Inclusion Criteria:

1. Must have metastatic breast cancer or locally advanced not amenable to curative therapy.
2. Measurable or evaluable disease are eligible.
3. Tumors must be Estrogen Receptor (ER)-positive and/or Progesterone Receptor (PR)-positive.
4. Human Epidermal Growth Factor Recepter 2 (HER2)-positive tumors are allowed but must have failed Herceptin therapy.
5. Postmenopausal
6. No more than 3 lines of chemotherapy
7. No more than 3 lines of hormonal therapy
8. Bisphosphonates may be given according to their product license
9. Left ventricular ejection fraction within institutional normal limits
10. Liver function and kidney function tests within the upper limit of normal. In patients with liver metastasis, liver function tests should be < 5 times the upper limit of normal.
11. Adequate blood counts
12. Normal thyroid function tests.
13. Patients with Central Nervous System (CNS) metastatic disease are allowed if the disease is stable for more than 3 months by CT or MRI.
14. Adequate general health (Eastern Cooperative Oncology Group (ECOG) performance status 0-2).
15. Able to give informed consent and follow the procedures of the study.

Exclusion Criteria:

1. Patients previously treated with exemestane in any setting.
2. Patients previously treated with sunitinib.
3. Patients with cardiac dysfunction or active cardiac disease
4. Patients with uncontrolled CNS metastasis.
5. Poorly controlled hypertension
6. Blood counts or liver and kidney tests that fall outside the ranges outlined in inclusion criteria 9-10 above.
7. ECOG performance status 3 or 4.
8. History of other malignancy within the last 5 years, except for carcinoma in situ of the cervix or basal cell carcinoma of the skin.
9. History of a cerebrovascular accident, non-catheter related deep vein thrombosis, or pulmonary embolism in the last 5 years.
10. Major surgical procedure or significant traumatic injury within 28 days prior to study entry.
11. Premenopausal status.
12. History of receiving any investigational treatment within 28 days of study medication initiation.
13. Current known infection.
14. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease; wound healing disorders; ulcers; or bone fractures).
15. Medical or psychiatric condition that in the opinion of the principal investigator impair their ability to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimiawi, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Lester and Sue Smith Breast Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exemestane Plus Sutent
Started | 4
Completed | 2 (2 patients were off study due to AE.)
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Exemestane Plus Sutent
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression in Weeks
Description: Time from the first day of treatment to date of progression in weeks
Time Frame: Medical evaluation every 4 weeks;The study does not have a fixed time frame for each participant. Duration of therapy depends on individule response, evidence of disease progression and tolerance
Population: 2 patients developed disease progression.
Measure: Mean (Full Range); unit: week
Groups:
- Exemestane Plus Sunitinib: All patients enrolled on the study will receive treatment as follows:
  1. Exemestane 25 mg by mouth every day.
  2. Sunitinib 37.5 mg by mouth every day.
Arm/Group | Exemestane Plus Sunitinib
Number analyzed (Participants) | 2
week | 11.1 [10.9 to 11.3]

2. Secondary Outcome: Obtain Assessments of Overall Response Rate, Clinical Benefit Rate, and Overall Survival
Time Frame: 5 years
Population: The study was terminated early before target accrual. 4 patients were enrolled and received treatment. 2 patients developed progression and 2 patients was drop-off the study due to adverse events.
Measure: Number; unit: paticipants
Groups:
- Exemestane Plus Sunitinib: This is a single arm study. All patients received Exemestane 25mg per day and Sunitinib 37.5 mg per day.
Arm/Group | Exemestane Plus Sunitinib
Number analyzed (Participants) | 4
paticipants | NA — The study was terminated early before target accrual and the secondary analyses were not conducted due to insufficient number of participants with events.

3. Secondary Outcome: Determine the Safety and Tolerability
Time Frame: 5 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Exemestane Plus Sunitinib
Number analyzed (Participants) | 4
Participants | NA — The study was terminated early before target accrual and the secondary analyses were not conducted due to insufficient number of participants.

4. Secondary Outcome: Study Molecular Changes in Tissue Biopsies, Circulating Tumor Cells, and Circulating Endothelial Cells
Time Frame: 5 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: cell
Arm/Group | Exemestane Plus Sunitinib
Number analyzed (Participants) | 4
cell | NA [NA to NA] — The study was terminated early before target accrual. No correlative study was performed.

ADVERSE EVENTS:
Time Frame: Medical evaluation every 4 weeks. The study does not have a fixed time frame for each participant. Duration of therapy depends on individule response, evidence of disease progression and tolerance.
Arm/Group | Exemestane Plus Sutent
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exemestane Plus Sutent (N=4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exemestane Plus Sutent (N=4)
leukopenia (Blood and lymphatic system disorders) | 4 (4)
Hypertension (Cardiac disorders) | 3 (4)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Mucositis/stomatitis (Gastrointestinal disorders) | 2 (2)
Ocular/Visual (Eye disorders) | 1 (1)
pain (General disorders) | 1 (2)
platelets (Blood and lymphatic system disorders) | 2 (2)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Thrombosis/embolism (Vascular disorders) | 1 (1)
Thyroid function, low (Endocrine disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes